CLINICAL TRIAL: NCT05147324
Title: Individualized Planned Eating Patterns to Improve Glycemic Management in Adolescents With Type 1 Diabetes: A Pilot Clinical Trial
Brief Title: "MyPlan" - Individualized Planned Eating Patterns for Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-1337; 1R21DK125033-01A1 (NIH)
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus, Type 1; Feeding Behavior; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "MyPlan" - Individualized Planned Eating Pattern (Experimental): All youth enrolled in the study will receive the 6-month MyPlan behavioral intervention. Youth and their guardian will be paired with a dietitian to individualize the eating pattern and receive support in setting and refining action plans focused on adhering to the five eating behavior goals that define the eating pattern.
  Interventions: Behavioral: "MyPlan" - Individualized Planned Eating Pattern

INTERVENTIONS:
Behavioral: "MyPlan" - Individualized Planned Eating Pattern — Sessions involve a structured behavior change counseling module derived from FLEX (NCT01286350), DASH-4-Teens (NCT00585832), and a Social Cognitive Theory and Transtheoretical Model informed conceptual framework, which uses education, motivation and self-efficacy enhancement, goal setting, and problem-solving skills training to initiate and sustain eating pattern adherence. Sessions support incremental progress towards meeting all five eating behavior goals by helping youth develop action plans, troubleshoot barriers to adherence, and refine action plans to improve adherence. Youth log in MyFitnessPal at least three days per week. Logs are used to assess and troubleshoot adherence, support youth in developing and refining action plans, and reward youth with points. Incentives are allocated using a point scheme designed to promote logging and goal achievement. Formal adjustment of the eating pattern is based on adherence according to logs and youth/guardian acceptability.
  Other Names: "MyPlan"

SUMMARY:
The purpose of this study is to test the acceptability and effectiveness of an individualized eating strategy as part of diabetes self-management to improve glycemic levels among youth with type 1 diabetes (T1D) and suboptimal glycemic management. Investigators will assess participant acceptability of and adherence to a 6-month individualized eating strategy ("MyPlan") characterized by approximate day-to-day consistency in the frequency and timing of meals and snacks and distribution of carbohydrate throughout the day. Within-individual change in glycemic levels between baseline and 6-months of the study will also be compared. The goal of the study is to inform the design of a future randomized clinical trial to test the addition of the MyPlan eating strategy to ongoing diabetes clinical care among youth with T1D.

DETAILED DESCRIPTION:
This is a pilot, single-arm clinical trial to assess whether "MyPlan" is an acceptable and effective dietary strategy to be included in future fully powered trials aimed at optimizing diabetes outcomes in youth with T1D. Youth and guardian dyads will be enrolled for a total of 6 months, during which time dyads will be counseled to follow an individualized eating pattern ("MyPlan") defined by five eating behavior goals: 3-4 meals per day and 1-2 optional snacks; eating occasions no less than 2 hours or greater than 4 hours apart; target carbohydrate ranges for each eating occasion; no post-dinner snacking; eating occasion within 1-2 hours of waking. The plan, including the eating behavior goals, will be tailored to youth and family routines and preferences. Registered dieticians will support participant adherence to the plan via telehealth counseling sessions on a weekly basis for the first 2 months followed by bi-weekly sessions for 4 months. Investigators will assess a) acceptability of the eating pattern and counseling strategy according to youth and guardians; b) youth adherence to the five eating behavior targets; c) change in youth glycemic levels between baseline and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Youth 12-17 years old
* History of T1D of at least one year
* HbA1c 7.5-11%
* Guardian willing to also participate
* English as preferred language

Exclusion Criteria:

* Youth with other metabolic disorders, unstable thyroid disease, diagnosed eating disorders, prohibitively strict dietary restrictions, or those with other serious condition that renders participation inappropriate.
* Females who are pregnant, breast feeding, planning to become pregnant during the study period or delivered a baby in the last 12 months.
* Unwillingness to follow a personalized eating plan for 6 months or complete MyFitnessPal logs at least 3 days/week throughout the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Mayer-Davis, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Sarah Couch, PhD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 36 months following publication. No end date.
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Writing Group for the DCCT/EDIC Research Group; Orchard TJ, Nathan DM, Zinman B, Cleary P, Brillon D, Backlund JY, Lachin JM. Association between 7 years of intensive treatment of type 1 diabetes and long-term mortality. JAMA. 2015 Jan 6;313(1):45-53. doi: 10.1001/jama.2014.16107. PMID 25562265
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Smart CE, Annan F, Bruno LP, Higgins LA, Acerini CL; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Nutritional management in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:135-53. doi: 10.1111/pedi.12175. No abstract available. PMID 25182313
- [Background] Weissberg-Benchell J, Glasgow AM, Tynan WD, Wirtz P, Turek J, Ward J. Adolescent diabetes management and mismanagement. Diabetes Care. 1995 Jan;18(1):77-82. doi: 10.2337/diacare.18.1.77. PMID 7698052
- [Background] Overby NC, Margeirsdottir HD, Brunborg C, Anderssen SA, Andersen LF, Dahl-Jorgensen K; Norwegian Study Group for Childhood Diabetes. Physical activity and overweight in children and adolescents using intensified insulin treatment. Pediatr Diabetes. 2009 Apr;10(2):135-41. doi: 10.1111/j.1399-5448.2008.00454.x. Epub 2008 Aug 20. PMID 18721165
- [Background] Overby NC, Margeirsdottir HD, Brunborg C, Andersen LF, Dahl-Jorgensen K. The influence of dietary intake and meal pattern on blood glucose control in children and adolescents using intensive insulin treatment. Diabetologia. 2007 Oct;50(10):2044-51. doi: 10.1007/s00125-007-0775-0. Epub 2007 Aug 9. PMID 17687538
- [Background] Li C, D'Agostino RB Jr, Dabelea D, Liese AD, Mayer-Davis EJ, Pate R, Merchant AT. Longitudinal association between eating frequency and hemoglobin A1c and serum lipids in diabetes in the SEARCH for Diabetes in Youth study. Pediatr Diabetes. 2018 Apr 30:10.1111/pedi.12690. doi: 10.1111/pedi.12690. Online ahead of print. PMID 29708292
- [Background] Wolever TM, Hamad S, Chiasson JL, Josse RG, Leiter LA, Rodger NW, Ross SA, Ryan EA. Day-to-day consistency in amount and source of carbohydrate intake associated with improved blood glucose control in type 1 diabetes. J Am Coll Nutr. 1999 Jun;18(3):242-7. doi: 10.1080/07315724.1999.10718858. PMID 10376780
- [Background] International Hypoglycaemia Study Group. Glucose Concentrations of Less Than 3.0 mmol/L (54 mg/dL) Should Be Reported in Clinical Trials: A Joint Position Statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2017 Jan;40(1):155-157. doi: 10.2337/dc16-2215. Epub 2016 Nov 21. No abstract available. PMID 27872155
- [Background] Beaton GH, Milner J, Corey P, McGuire V, Cousins M, Stewart E, de Ramos M, Hewitt D, Grambsch PV, Kassim N, Little JA. Sources of variance in 24-hour dietary recall data: implications for nutrition study design and interpretation. Am J Clin Nutr. 1979 Dec;32(12):2546-59. doi: 10.1093/ajcn/32.12.2546. No abstract available. PMID 506977
- [Background] Posner BM, Smigelski C, Duggal A, Morgan JL, Cobb J, Cupples LA. Validation of two-dimensional models for estimation of portion size in nutrition research. J Am Diet Assoc. 1992 Jun;92(6):738-41. No abstract available. PMID 1607574
- [Background] Kozey Keadle S, Lyden K, Hickey A, Ray EL, Fowke JH, Freedson PS, Matthews CE. Validation of a previous day recall for measuring the location and purpose of active and sedentary behaviors compared to direct observation. Int J Behav Nutr Phys Act. 2014 Feb 3;11:12. doi: 10.1186/1479-5868-11-12. PMID 24490619
- [Background] Clark BK, Pavey TG, Lim RF, Gomersall SR, Brown WJ. Past-day recall of sedentary time: Validity of a self-reported measure of sedentary time in a university population. J Sci Med Sport. 2016 Mar;19(3):237-241. doi: 10.1016/j.jsams.2015.02.001. Epub 2015 Feb 21. PMID 25766507
- [Background] Maahs DM, Mayer-Davis E, Bishop FK, Wang L, Mangan M, McMurray RG. Outpatient assessment of determinants of glucose excursions in adolescents with type 1 diabetes: proof of concept. Diabetes Technol Ther. 2012 Aug;14(8):658-64. doi: 10.1089/dia.2012.0053. PMID 22853720
- [Background] Markowitz JT, Butler DA, Volkening LK, Antisdel JE, Anderson BJ, Laffel LM. Brief screening tool for disordered eating in diabetes: internal consistency and external validity in a contemporary sample of pediatric patients with type 1 diabetes. Diabetes Care. 2010 Mar;33(3):495-500. doi: 10.2337/dc09-1890. Epub 2009 Dec 23. PMID 20032278
- [Background] Couch SC, Saelens BE, Levin L, Dart K, Falciglia G, Daniels SR. The efficacy of a clinic-based behavioral nutrition intervention emphasizing a DASH-type diet for adolescents with elevated blood pressure. J Pediatr. 2008 Apr;152(4):494-501. doi: 10.1016/j.jpeds.2007.09.022. Epub 2007 Nov 5. PMID 18346503
- [Background] Kichler JC, Seid M, Crandell J, Maahs DM, Bishop FK, Driscoll KA, Standiford D, Hunter CM, Mayer-Davis E. The Flexible Lifestyle Empowering Change (FLEX) intervention for self-management in adolescents with type 1 diabetes: Trial design and baseline characteristics. Contemp Clin Trials. 2018 Mar;66:64-73. doi: 10.1016/j.cct.2017.12.006. Epub 2017 Dec 24. PMID 29277316
- [Background] Mayer-Davis EJ, Maahs DM, Seid M, Crandell J, Bishop FK, Driscoll KA, Hunter CM, Kichler JC, Standiford D, Thomas JM; FLEX Study Group. Efficacy of the Flexible Lifestyles Empowering Change intervention on metabolic and psychosocial outcomes in adolescents with type 1 diabetes (FLEX): a randomised controlled trial. Lancet Child Adolesc Health. 2018 Sep;2(9):635-646. doi: 10.1016/S2352-4642(18)30208-6. Epub 2018 Jul 30. PMID 30119757

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-two guardians and youth were enrolled as dyads. A total of 44 dyads were included in the analysis.
Groups:
- "MyPlan" - Individualized Eating Pattern: All youth enrolled in the study will receive the 6-month MyPlan behavioral intervention. Youth will be paired with a dietitian to individualize the eating plan and receive support in setting and refining action plans focused on adhering to the five eating behavior goals that define the eating plan.
  "MyPlan" - Individualized Eating Pattern: Sessions involve a structured behavior change counseling module derived from FLEX (NCT01286350), DASH-4-Teens (NCT00585832), and a Social Cognitive Theory and Transtheoretical Model informed conceptual framework, which uses education, motivation and self-efficacy enhancement, goal setting, and problem-solving skills training to initiate and sustain eating plan adherence. Sessions support incremental progress towards meeting all five eating behavior goals by helping youth develop action plans, troubleshoot barriers to adherence, and refine action plans to improve adherence. Youth log in MyFitnessPal three days per week. Logs are used to assess and troubleshoot adherence, support youth in developing and refining action plans, and reward youth with points. Incentives are allocated using a point scheme designed to promote logging and goal achievement. Formal adjustment of eating plan at three months is based on weight status, adherence according to logs, and youth/guardian acceptability.
Period: Overall Study
Arm/Group | "MyPlan" - Individualized Eating Pattern
Started (Number Started reflects dyad pairs (i.e., 52 Guardians + 52 Youth).) | 52
Completed (Number Completed reflects dyad pairs (i.e., 44 Guardians + 44 Youth).) | 44
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Baseline data was only collected for youth.
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 30
  Non-Hispanic Black | 9
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent Time in Range (Baseline)
Description: Percentage of time spent in the glycemic range of 70-180 mg/dL between Baseline week 0-2 week of blinded continuous glucose monitor (CGM) wear time.
Time Frame: Baseline (Week 0-2)
Population: Data from study-provided continuous glucose monitors was not available for 10 participants.
Measure: Mean (Standard Deviation); unit: percentage of CGM wear time
Arm/Group | "MyPlan" - Individualized Planned Eating Pattern
Number analyzed (Participants) | 34
percentage of CGM wear time | 40.6 (3.1)
Statistical Analysis 1: Comparison: "MyPlan" - Individualized Planned Eating Pattern; Test type: Superiority; p = 0.70, t-test, 2 sided

2. Primary Outcome: Percent Time in Range (Week 22-24)
Description: Percentage of time spent in the glycemic range of 70-180 mg/dL during Week 22-24 of blinded continuous glucose monitor (CGM) wear time.
Time Frame: Week 22-24
Population: Data from study-provided continuous glucose monitors was not available for 7 participants.
Measure: Mean (Standard Deviation); unit: percentage of CGM wear time
Arm/Group | "MyPlan" - Individualized Planned Eating Pattern
Number analyzed (Participants) | 37
percentage of CGM wear time | 41.7 (2.4)
Statistical Analysis 1: Comparison: "MyPlan" - Individualized Planned Eating Pattern; Test type: Superiority; p = 0.70, t-test, 2 sided

3. Primary Outcome: Adherence to Each Eating Behavior Goal
Description: Percentage of participants who adhered to each eating behavior goal assessed through two unannounced 24-hour dietary recalls (1 weekday and 1 weekend day) collected during Week 22-24:
  Goal 1. 3-4 meals and 0-2 snacks; Goal 2. Spacing of meals/snacks >2 hours and <4 hours apart; Goal 3. Carbohydrate gram target ranges at meals (>15% daily carbohydrate) and snacks; Goal 4. No snacking after dinner; Goal 5. Meal/snack consumed ≤2 hours of waking;
Time Frame: Between Week 22 and Week 24
Population: Data are reported for a total of 41 unique participants between weekday and weekend 24-hour dietary recall. Neither a weekday nor weekend day 24-hour dietary recall was completed for 3 participants. Of the 41 participants, one did not complete a weekday 24-hour dietary recall and 3 participants did not complete a weekend 24-hour dietary recall.
Measure: Number; unit: percentage of participants
Arm/Group | "MyPlan" - Individualized Planned Eating Pattern
Number analyzed (Participants) | 41
percentage of participants
  Goal 1 Weekday: number analyzed (Participants) | 40
  Goal 1 Weekday | 92.5
  Goal 2 Weekday: number analyzed (Participants) | 40
  Goal 2 Weekday | 30.0
  Goal 3 Weekday: number analyzed (Participants) | 40
  Goal 3 Weekday | 87.5
  Goal 4 Weekday: number analyzed (Participants) | 40
  Goal 4 Weekday | 75.0
  Goal 5 Weekday: number analyzed (Participants) | 40
  Goal 5 Weekday | 92.5
  Goal 1 Weekend: number analyzed (Participants) | 38
  Goal 1 Weekend | 81.6
  Goal 2 Weekend: number analyzed (Participants) | 38
  Goal 2 Weekend | 36.8
  Goal 3 Weekend: number analyzed (Participants) | 38
  Goal 3 Weekend | 86.8
  Goal 4 Weekend: number analyzed (Participants) | 38
  Goal 4 Weekend | 76.3
  Goal 5 Weekend: number analyzed (Participants) | 38
  Goal 5 Weekend | 94.7

4. Primary Outcome: Adherence to 0-5 Eating Behavior Goals
Description: Percentage of participants who adhered to 0-5 eating behavior goals assessed through two unannounced 24-hour dietary recalls (1 weekday and 1 weekend day) collected during Week 22 - 24.
  Goal 1. 3-4 meals and 0-2 snacks; Goal 2. Spacing of meals/snacks >2 hours and <4 hours apart Goal 3. Carbohydrate gram target ranges at meals (>15% daily carbohydrate) and snacks Goal 4. No snacking after dinner Goal 5. Meal/snack consumed ≤2 hours of waking
Time Frame: Between Week 22 and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | "MyPlan" - Individualized Planned Eating Pattern
Number analyzed (Participants) | 41
percentage of participants
  Adherent to 0 Goals Weekday: number analyzed (Participants) | 40
  Adherent to 0 Goals Weekday | 0.0
  Adherent to 1 Goal Weekday: number analyzed (Participants) | 40
  Adherent to 1 Goal Weekday | 0.0
  Adherent to 2 Goals Weekday: number analyzed (Participants) | 40
  Adherent to 2 Goals Weekday | 7.5
  Adherent to 3 Goals Weekday: number analyzed (Participants) | 40
  Adherent to 3 Goals Weekday | 25.0
  Adherent to 4 Goals Weekday: number analyzed (Participants) | 40
  Adherent to 4 Goals Weekday | 50.0
  Adherent to 5 Goals Weekday: number analyzed (Participants) | 40
  Adherent to 5 Goals Weekday | 17.5
  Adherent to 0 Goals Weekend: number analyzed (Participants) | 38
  Adherent to 0 Goals Weekend | 0.0
  Adherent to 1 Goal Weekend: number analyzed (Participants) | 38
  Adherent to 1 Goal Weekend | 0.0
  Adherent to 2 Goals Weekend: number analyzed (Participants) | 38
  Adherent to 2 Goals Weekend | 7.9
  Adherent to 3 Goals Weekend: number analyzed (Participants) | 38
  Adherent to 3 Goals Weekend | 21.1
  Adherent to 4 Goals Weekend: number analyzed (Participants) | 38
  Adherent to 4 Goals Weekend | 58.9
  Adherent to 5 Goals Weekend: number analyzed (Participants) | 38
  Adherent to 5 Goals Weekend | 13.2

5. Primary Outcome: Mean Adherence to Overall Eating Behavior Pattern
Description: Mean number of eating behavior goals (range: 0-5) adhered to by participants as assessed through two unannounced 24-hour dietary recalls (1 weekday and 1 weekend day) collected during Week 22 - 24:
  Goal 1. 3-4 meals and 0-2 snacks; Goal 2. Spacing of meals/snacks >2 hours and <4 hours apart; Goal 3. Carbohydrate gram target ranges at meals (>15% daily carbohydrate) and snacks; Goal 4. No snacking after dinner; Goal 5. Meal/snack consumed ≤2 hours of waking;
Time Frame: Between Week 22 and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: goals
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 41
goals
  Number of Goals - Weekday: number analyzed (Participants) | 40
  Number of Goals - Weekday | 3.8 (0.83)
  Number of Goals - Weekend: number analyzed (Participants) | 38
  Number of Goals - Weekend | 4.0 (0.80)

6. Primary Outcome: Mean Acceptability Score (Youth)
Description: Mean composite acceptability score (range: 5-20) calculated from Likert responses (1- Strongly Agree, 2- Agree, 3- Disagree, 4- Strongly Disagree) to 5 items from an instrument that captures ease of eating pattern adoption, satisfaction, food enjoyment, sustainability, and ease of blood sugar management as perceived by youth. Lower composite acceptability scores indicate greater acceptability (5 - highly acceptable 20 - highly unacceptable).
Time Frame: Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 44
score on a scale | 7.8 (2.4)

7. Primary Outcome: Acceptability Percentage (Youth)
Description: Percentage of youth with a mean acceptability score (range: 5-20) <=10. Lower acceptability scores indicate greater acceptability (5 - highly acceptable 20 - highly unacceptable) where a score >10 indicates the eating pattern is unacceptable. Scores calculated from Likert responses (1- Strongly Agree 2- Agree 3- Disagree 4- Strongly Disagree) to 5 scored items from an instrument that captures ease of eating pattern adoption, satisfaction, food enjoyment, sustainability, and ease of blood sugar management as perceived by youth.
Time Frame: Week 26
Measure: Number; unit: percentage of participants
Arm/Group | "MyPlan" - Individualized Planned Eating Pattern
Number analyzed (Participants) | 44
percentage of participants | 86.4

8. Primary Outcome: Mean Acceptability Score (Guardian)
Description: Mean composite acceptability score (range: 5-20) calculated from Likert responses (1- Strongly Agree, 2- Agree, 3- Disagree, 4- Strongly Disagree) to 5 items from an instrument that captures ease of eating pattern adoption, satisfaction, food enjoyment, sustainability, and ease of blood sugar management as perceived by youth's guardian. Lower composite acceptability scores indicate greater acceptability (5 - highly acceptable 20 - highly unacceptable).
Time Frame: Week 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 44
score on a scale | 7.8 (2.3)

9. Primary Outcome: Acceptability Percentage (Guardian)
Description: Percentage of guardians with a mean acceptability score (range: 5-20) <=10. Lower acceptability scores indicate greater acceptability (5 - highly acceptable 20 - highly unacceptable) where a score >10 indicates the eating pattern is unacceptable. Scores calculated from Likert responses (1- Strongly Agree 2- Agree 3- Disagree 4- Strongly Disagree) to 5 scored items from an instrument that captures ease of eating pattern adoption, satisfaction, food enjoyment, sustainability, and ease of blood sugar management as perceived by youth's guardian.
Time Frame: Week 26
Measure: Number; unit: percentage of guardians
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 44
percentage of guardians | 93.2

10. Secondary Outcome: Change in Hemoglobin A1c Percentage
Description: Change in point-of-care hemoglobin A1c (HbA1c) percentage.
Time Frame: Baseline (Week 0) and Endline (Week 26)
Population: HbA1c was not completed for the endline visit at Week 26 for 3 participants who completed this visit remotely.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | "MyPlan" - Individualized Eating Pattern
Number analyzed (Participants) | 41
percentage of red blood cells | -0.32 (0.89)
Statistical Analysis 1: Comparison: "MyPlan" - Individualized Eating Pattern; Test type: Superiority; p = 0.03, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, up to approximately 26 weeks.
Description: Adverse events were not collected for Guardians.
Arm/Group | "MyPlan" - Individualized Eating Pattern
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT05147324/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT05147324/ICF_000.pdf